CLINICAL TRIAL: NCT00654758
Title: A Phase 1b Trial to Evaluate the Safety and Pharmacokinetics of Volociximab (M200) in Combination With Carboplatin and Paclitaxel in Subjects With Previously Untreated Stage IIIB/IV Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Phase 1b Study With Volociximab in Combination With Carboplatin and Paclitaxel in First-line, Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M200-1211; 2007-003396-39 (EudraCT Number)
Record Dates: First submitted 2008-04-04; First posted 2008-04-09 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2012-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: cancer; carcinoma; chemotherapy; monoclonal antibody therapy; anti-angiogenesis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Carcinoma | interventions — volociximab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Escalating doses of volociximab at 10, 20, and 30 (or 15) mg/kg with carboplatin and paclitaxel.
  Interventions: Drug: M200 (Volociximab), Carboplatin, Paclitaxel

INTERVENTIONS:
Drug: M200 (Volociximab), Carboplatin, Paclitaxel — Volociximab will be administered via IV infusion at 10, 20, and 15 or 30 mg/kg with an additional loading dose in the 10, 20, and 15 mg/kg dose levels during the first cycle. Volociximab will be given for at least 6 cycles (3 weeks/cycle) and subjects who have stable disease at the end of 6 cycles may continue to receive volociximab alone until disease progression. Carboplatin is administered via IV infusion and dosed based on the Calvert formula (with a target area AUC of 6 mg/mL/min) for up to 6 cycles (3 weeks/cycle). Paclitaxel is administered via IV infusion and dosed at 200 mg/m2 for up to 6 cycles (3 weeks/cycle). All three drugs, when given in combination, will be infused on the same day in the following sequence: volociximab, paclitaxel, carboplatin.
  Other Names: Volociximab (M200)

SUMMARY:
The primary purpose of this study is to examine the safety of volociximab in combination with a standard treatment of carboplatin and paclitaxel in subjects previously untreated with chemotherapy for advanced stage (IIIB/IV) non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This Phase 1b, multicenter, open-label, dose-escalation study will evaluate the safety and pharmacokinetics (PK) of volociximab in combination with carboplatin and paclitaxel (C/P) as first-line treatment in subjects with Stage IIIB or IV non-small cell lung cancer (NSCLC). Volociximab doses of 10, 20, and 30 mg/kg (or 15 mg/kg if 20 mg/kg is not tolerable) with carboplatin/paclitaxel chemotherapy will be tested for determining the maximum tolerated dose (MTD). Subjects will be dosed once very 3 weeks for up to 6 cycles.

Volociximab is a high-affinity, chimeric monoclonal antibody that specifically binds to α5β1 integrin, a cell-surface receptor for fibronectin. Volociximab blocks the binding of α5β1 to fibronectin, thereby inhibiting a pivotal interaction required for angiogenesis.

More than 170 subjects with various solid tumor types have received volociximab in Phase 1 and Phase 2 single and combination studies. At the doses tested, there has not been a dose limiting toxicity (DLT) or a maximum tolerated dose (MTD) defined.

ELIGIBILITY:
Inclusion Criteria

1. Males and females at least 18 years of age.
2. Stage IIIB or IV or recurrent NSCLC.
3. Measurable and/or evaluable disease according to RECIST.
4. No prior chemotherapy, biological therapy or immunotherapy for Stage IIIB/IV disease. Adjuvant therapy for early stage disease must have been completed > or = 6 months prior to Cycle 1, Day 1 of this study.
5. Eastern Cooperative Oncology Group (ECOG) performance status < or =1.
6. A negative pregnancy test (serum or urine) in women of childbearing potential at screening.

Exclusion Criteria

1. Known allergy or sensitivity to murine proteins, chimeric antibodies or other components of the product, Cremophor EL (polyoxyethylated castor oil), cisplatin, or other platinum-containing compounds.
2. Absolute neutrophil count (ANC) <1500/mm3, hemoglobin level <9 g/dL, or a platelet count <100,000/mm3.
3. Aspartate transaminase (AST), alanine transaminase (ALT), or alkaline phosphatase values of .2.5 of the upper limits of normal values (ULN) (>5 ULN for subjects with liver metastases) or alkaline phosphatase values >2.5 ULN (unless documented bone metastases are responsible for the increase of alkaline phosphatase); total bilirubin >1.5 mg/dL, or serum creatinine >1.8 mg/dL.
4. Radiation therapy within 1 month before Cycle 1, Day 1.
5. Documented symptomatic central nervous system (CNS) tumor or CNS metastases.
6. History of thromboembolic events, including cardiovascular or cerebrovascular events (ie, acute myocardial infarction [AMI], stroke) within 1 year prior to Cycle 1, Day 1.
7. History of known bleeding disorders and coagulation defects.
8. History of significant hemoptysis (ie, > or =1/2 teaspoon red blood per event) or gastrointestinal bleeding within 1 year prior to Cycle 1, Day 1.
9. Major surgery (eg, exploratory laparotomy) within 4 weeks prior to Cycle 1, Day 1 of the study.
10. Clinically significant or unstable medical conditions including, but not limited to, uncontrolled diabetes mellitus requiring insulin, uncontrolled hypertension, or uncontrolled or symptomatic orthostatic hypotension.
11. Oxygen-dependent chronic obstructive pulmonary disease.
12. Known active infections requiring intravenous (IV) antibiotics, antivirals, or antifungals, including but not limited to chronic human immunodeficiency virus, hepatitis B, or hepatitis C infection.
13. Prior bone marrow or stem cell transplant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of volociximab given at different doses in combination with carboplatin and paclitaxel | Dose escalation phase of the trial

SECONDARY OUTCOMES:
Pharmacokinetics of volociximab | Approximately 2.5 years
Efficacy of volociximab in combination with carboplatin/paclitaxel | Approximately 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mihail Obrocea, MD, Study Director — Abbott

REFERENCES:
- [Result] Besse B, Tsao LC, Chao DT, Fang Y, Soria JC, Almokadem S, Belani CP. Phase Ib safety and pharmacokinetic study of volociximab, an anti-alpha5beta1 integrin antibody, in combination with carboplatin and paclitaxel in advanced non-small-cell lung cancer. Ann Oncol. 2013 Jan;24(1):90-6. doi: 10.1093/annonc/mds281. Epub 2012 Aug 16. PMID 22904239